CLINICAL TRIAL: NCT03549793
Title: Can Dance Therapy Improve Motor Learning in Parkinson's Disease?
Brief Title: Can Dance Therapy Improve Motor Learning in Parkinson's Disease (PD)?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dance therapy in PD
Record Dates: First submitted 2018-05-07; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Dance Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to experimental group or control group. Both of the groups undergo a rehabilitation treatment. The experimental group undergoes 4-week MIRT (Multidisciplinary Intensive Rehabilitation Treatment) + dance therapy. The control group undergoes 4-week MIRT (Multidisciplinary Intensive Rehabilitation Treatment) + exercises
Who Masked: Investigator
Masking Description: The investigator are neurologists, blinded to the treatment received by the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dance thrapy (Experimental): 4-week Multidisciplinary Rehabilitation Treatment + Dance Therapy Treatment (2 hours par week)
  Interventions: Behavioral: Dance Therapy
- exercises without dance (Active Comparator): 4-week Multidisciplinary Rehabilitation Treatment + Exercises without music (2 hours par week)
  Interventions: Behavioral: exercises without dance

INTERVENTIONS:
Behavioral: Dance Therapy — the intervention is aimed to ameliorate, through dancing, crucial motor symptoms in PD patients, as walking, balance, postural changes and arm swing
  Arms: dance thrapy
Behavioral: exercises without dance — the intervention consists of exercises aimed at training the walking, the balance, the postural changes and the arm swing
  Arms: exercises without dance

SUMMARY:
In order to find the most effective rehabilitative therapies for Parkinsonian patients, the present study is aimed to evaluate whether, in a multidisciplinary intensive rehabilitation treatment, the dance therapy, applied to the motor learning, promote additional benefits.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2.5-3 according to the Hoehn and Yahr scale (H&Y);
* Stable pharmacological treatment for the last 6 weeks before the enrolment and during the hospitalization;

Exclusion Criteria:

* Any focal brain lesion detected in brain imaging studies (CT or MRI) performed in the previous 12 months;
* Drug-induced dyskinesias;
* Disturbing resting and/or action tremor, corresponding to scores 2-4 in the specific items of UPDRS III;
* Behavioral disturbances (evaluated with Neuropsychiatric Inventory);
* Visual and auditory dysfunctions according to the general clinical evaluation and medical history;
* cognitive decline (MMSE correct score < 24)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test (TUG) | 4 weeks
  To determine fall risk and measure the progress of balance, sit to stand, and walking.

SECONDARY OUTCOMES:
6 Minutes Walking Test (6MWT) | 4 weeks
  The 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Balance Berg Scale (BBS) | 4 weeks
  to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.

OTHER OUTCOMES:
delayed recall of items | 4 weeks
  number of specific items correctly performed in recall phase

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Department of Parkinson's disease, Movement Disorders and Brain Injury Rehabilitation, "Moriggia-Pelascini" Hospital - Via Pelascini, 3, 22015, Gravedona ed Uniti, Como, Italy
Locations (1):
- Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No